CLINICAL TRIAL: NCT00398866
Title: A Study of Hyaluronan (Synvisc) for the Treatment of Osteoarthritis in the Thumb: Randomized Control Trial
Brief Title: A Study of Hyaluronan for the Treatment of Osteoarthritis in the Thumb
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: K23AR050607 (NIH); K23AR050607 (NIH); 5K23AR050607-04 (NIH); 26043 (Other: HSS IRB)
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Results first posted 2017-07-07 (Actual); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Osteoarthritis
Keywords: Hyaluronan; Carpometacarpal; Outcomes; Carpometacarpal Joints
MeSH Terms: conditions — Osteoarthritis | interventions — hylan; Hyaluronic Acid; Anesthesia, Local; Triamcinolone Acetonide; Triamcinolone; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Bupivicaine (local anesthetic)
  Interventions: Drug: Bupivicaine (local anesthesia injection)
- 2 (Active Comparator): Corticosteroid (trimcinolone (Kenalog) 40 mg)
  Interventions: Drug: Kenalog (triamcinolone; corticosteroid injection)
- 3 (Experimental): Synvisc
  Interventions: Drug: Synvisc (Hylan G-F20; hyaluronan injection)

INTERVENTIONS:
Drug: Synvisc (Hylan G-F20; hyaluronan injection) — 1 ml of hyaluronan (Synvisc) injected once a week for 2 consecutive weeks
  Other Names: Synvisc, Hyalgan, Hyaluronic Acid
  Arms: 3
Drug: Bupivicaine (local anesthesia injection) — 1 ml of bupivicaine 0.5% injected once a week for 2 weeks
  Arms: 1
Drug: Kenalog (triamcinolone; corticosteroid injection) — 1 ml (40mg) of triamcinolone (Kenalog) injected the first week, followed by a placebo injection of 1 ml 0.5% bupivacaine the second week; Kenalog is a non-suspension steroid preparation and is less likely to cause post-injection flares than a suspension preparation
  Arms: 2

SUMMARY:
Hyaluronan is a man-made preparation of a protein complex that occurs naturally in joints and that is often low in people with osteoarthritis. Although hyaluronan has been used in millions of people with knee osteoarthritis, it is not yet FDA approved for use in the thumb. The purpose of this study is to determine the safety and effectiveness of hyaluronan in relieving arthritis symptoms at the base of the thumb and to compare it to corticosteroids and local anesthetic.

The principle hypothesis is that treating osteoarthritis at the carpometacarpophalangeal (CMC) joint with injectable hyaluronan will results in greater pain relief, higher patient satisfaction, and better functional outcomes than treating with placebo injections (local anesthetic) or with corticosteroid injections. Treating CMC osteoarthritis with corticosteroid injections will result in greater pain relief, higher patient satisfaction, and better functional outcomes than treating with placebo injections. Patients with worse pre-treatment function will have less improvement and worse post-treatment results after administration of corticosteroid or hyaluronan.

DETAILED DESCRIPTION:
Osteoarthritis involves a wearing down of the cartilage within a joint. It can affect any joint in the body, but it most commonly affects joints in the hands, hips, knees, and spine. Over the last few years, a new medicine called hyaluronan has been used for treating osteoarthritis. Hyaluronan is a man-made preparation of a protein complex that occurs naturally in joints and that is often low in people with osteoarthritis. Although hyaluronan has been used in millions of people with knee osteoarthritis, it is not yet FDA approved for use in the thumb. The purpose of this study is to determine the safety and effectiveness of hyaluronan in relieving arthritis symptoms at the base of the thumb and to compare it to corticosteroids and local anesthetic. Specifically, the study will evaluate pain relief, patient satisfaction, and functional outcomes among participants.

Participation in this study will last 26 weeks. Screening will include a questionnaire and an x-ray of the affected thumb. Eligible participants will then be randomly assigned to one of three treatments: two hyaluronan injections, one corticosteroid injection plus one local anesthetic injection, or two local anesthetic injections. Participants will receive the injections at the base of their thumb, and the first injection will be followed by the second injection a week later. There will be five study visits that will occur at baseline and Weeks 2, 4, 12, and 26. All study visits will include questionnaires, and except for the Week 2 study visit, they will also include an examination and evaluation of the affected thumb. Photographs of the thumb will be taken at baseline. The injections will occur at baseline and Week 2. At Weeks 8 and 20, questionnaires will be mailed to participants for them to complete. Upon completing the study, participants will have the option of receiving continued treatment with another round of hyaluronic injections.

ELIGIBILITY:
Inclusion Criteria:

* Presence of osteophytes or sclerosis at the carpometacarpal (CMC) joint
* Complaint of unacceptable pain despite modification of activity and a therapeutic dose of nonsteroidal anti-inflammatory drugs (NSAIDS), if tolerated
* If bilateral disease, only the most severely involved hand (as defined by the visual analog scale [VAS] for pain) will be entered in the study
* Able to follow instructions and complete questionnaires
* Failed conservative therapy with NSAIDS or COX-2 inhibitors
* Unable to tolerate COX-2 inhibitors

Exclusion Criteria:

* Previous traumatic dislocation, ligament tear, or fracture of the thumb in the affected hand
* Previous hand surgery on the affected hand
* Known hand comorbidities (e.g., active carpal tunnel syndrome, de Quervains tenosynovitis, etc.)
* Systemic rheumatic disease
* Bleeding diatheses or anti-coagulation
* Allergies to steroids, chicken products, bupivicaine, or adhesive (e.g., double-sided tape)
* Current use of oral or intravenous steroids
* Active systemic malignancies
* Hyaluronan injection in the target CMC joint in the last 6 months
* Steroid or hyaluronan injection in any other joint in the last 6 months
* Insulin dependent diabetes mellitus (IDDM)
* Active infection
* Pain in the index joint that is more than 40 out of 100 on a VAS Pain scale
* End Stage CMC osteoarthritis, equivalent to bone on bone, Kellgren and Lawrence Stage IV
* Grade 3 or 4 Eaton and Litter (E+L) Classification
* E+L 3: Advanced joint distraction, subchondral cysts, and sclerosis
* E+L 4: Involvement of several joint surfaces

Ages: 45 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-08; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Mandl, MD, MPH, Principal Investigator — Hospital for Special Surgery, New York
Locations (1):
- Hospital for Special Surgery, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the practices of Hospital for Special Surgery (HSS) physicians or were or self-referred. Study information was posted on the HSS website, clinicaltrials.gov, Craig's List and local newspapers. Recruitment occurred between 05/25/2007 and 07/15/2009.
Pre-assignment Details: 396 subjects screened 169 did not meet eligibility criteria 27 declined injection 200 subjects randomized
Groups:
- Bupivicaine: Bupivicaine (local anesthetic)
  Bupivicaine (local anesthesia injection): 1 ml of bupivicaine 0.5% injected once a week for 2 weeks
- Triamcinolone: Corticosteroid (triamcinolone (Kenalog) 40 mg)
  Kenalog (triamcinolone; corticosteroid injection): 1 ml (40mg) of triamcinolone (Kenalog) injected the first week, followed by a placebo injection of 1 ml 0.5% bupivacaine the second week; Kenalog is a non-suspension steroid preparation and is less likely to cause post-injection flares than a suspension preparation
- Hylan G-F 20: Synvisc
  Synvisc (Hylan G-F20; hyaluronan injection): 1 ml of hyaluronan (Synvisc) injected once a week for 2 consecutive weeks
Period: Overall Study
Arm/Group | Bupivicaine | Triamcinolone | Hylan G-F 20
Started | 66 | 68 | 66
Completed | 52 | 60 | 58
Not Completed | 14 | 8 | 8
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Lost to Follow-up | 7 | 6 | 4
Not completed — Withdrawal by Subject | 5 | 1 | 2
Not completed — Unable to complete requirements of study | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Triamcinolone: Corticosteroid (trimcinolone (Kenalog) 40 mg)
  Kenalog (triamcinolone; corticosteroid injection): 1 ml (40mg) of triamcinolone (Kenalog) injected the first week, followed by a placebo injection of 1 ml 0.5% bupivacaine the second week; Kenalog is a non-suspension steroid preparation and is less likely to cause post-injection flares than a suspension preparation
- Total: Total of all reporting groups
Arm/Group | Bupivicaine | Triamcinolone | Hylan G-F 20 | Total
Number analyzed (Participants) | 66 | 68 | 66 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.3 (9.3) | 66.6 (8.4) | 67.1 (10.1) | 66.7 (9.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender: Female | 50 | 40 | 45 | 135
  Gender: Male | 16 | 28 | 20 | 64
  Gender: No data | 0 | 0 | 1 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 58 | 61 | 61 | 180
  Race: Other | 8 | 7 | 4 | 19
  Race: No data | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Visual Analogue Scale (VAS)
Description: Pain intensity measured on a Visual Analog Scale with scores ranging from 0 to 100, with 100 = severe pain.
Time Frame: Baseline, 26 Weeks
Population: Patients who completed follow-up through 26 weeks
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Bupivicaine | Triamcinolone | Hylan G-F 20
Number analyzed (Participants) | 61 | 65 | 62
Units on a scale
  Pain VAS at Baseline | 57.1 (20.1) | 63.2 (20.2) | 60.7 (19.3)
  Pain VAS at 26 weeks | 42.9 (26.5) | 50.1 (29.4) | 49.8 (26.3)

2. Secondary Outcome: Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire
Description: Disabilities of the Arm, Shoulder and Hand (DASH) Questionnaire measures degree of disability on a scale of 0 to 100, with a higher score indicating greater disability.
Time Frame: Baseline, 26 Weeks
Population: Patients who completed follow-up through 26 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivicaine | Triamcinolone | Hylan G-F 20
Number analyzed (Participants) | 61 | 65 | 62
units on a scale
  DASH at Baseline | 25.7 (17.1) | 28.9 (17.9) | 28.8 (17.3)
  Dash at 26 Weeks | 24.2 (17.4) | 27.0 (18.0) | 26.1 (19.0)

ADVERSE EVENTS:
Arm/Group | Bupivicaine | Triamcinolone | Hylan G-F 20
Serious Adverse Events (participants affected / at risk) | 1/66 | 0/68 | 2/66
Other Adverse Events (participants affected / at risk) | 2/66 | 10/68 | 3/66
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivicaine (N=66) | Triamcinolone (N=68) | Hylan G-F 20 (N=66)
Fall--hand injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Emergency Cholecystecomy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mitral Valve Surgery (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivicaine (N=66) | Triamcinolone (N=68) | Hylan G-F 20 (N=66)
Skin Atrophy or Depigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 0 (0)
Pain, Swelling, or Numbness in Hand (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (3) | 2 (2)
Skin and Nail Abnormalities (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Positive ANA Test (Previous status unknown) (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No